CLINICAL TRIAL: NCT06735235
Title: Evaluation of Salivary Fluoride Clearance Following the Use of Three MFP-Containing Dentifrices
Brief Title: Salivary Fluoride Clearance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2021061
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Period 1 (Other): 0 ppm F (placebo, negative control), 250 ppm F as MFP (dose-response control), 1100 ppm F as MFP (reference), 2800 ppm F as MFP (dose-response control)
  Interventions: Drug: 0 ppm F; Drug: 250 ppm F as MFP; Drug: 1100 ppm as MFP; Drug: 2800 ppm F as MFP
- Period 2 (Other): 0 ppm F (placebo, negative control), 250 ppm F as MFP (dose-response control), 1100 ppm F as MFP (reference), 2800 ppm F as MFP (dose-response control)
  Interventions: Drug: 0 ppm F; Drug: 250 ppm F as MFP; Drug: 1100 ppm as MFP; Drug: 2800 ppm F as MFP
- Period 3 (Other): 0 ppm F (placebo, negative control), 250 ppm F as MFP (dose-response control), 1100 ppm F as MFP (reference), 2800 ppm F as MFP (dose-response control)
  Interventions: Drug: 0 ppm F; Drug: 250 ppm F as MFP; Drug: 1100 ppm as MFP; Drug: 2800 ppm F as MFP
- Period 4 (Other): 0 ppm F (placebo, negative control), 250 ppm F as MFP (dose-response control), 1100 ppm F as MFP (reference), 2800 ppm F as MFP (dose-response control)
  Interventions: Drug: 0 ppm F; Drug: 250 ppm F as MFP; Drug: 1100 ppm as MFP; Drug: 2800 ppm F as MFP

INTERVENTIONS:
Drug: 0 ppm F — Each subject will be randomly assigned to this treatment during one of the four periods for this crossover study.
Drug: 250 ppm F as MFP — Each subject will be randomly assigned to this treatment during one of the four periods for this crossover study.
Drug: 1100 ppm as MFP — Each subject will be randomly assigned to this treatment during one of the four periods for this crossover study.
Drug: 2800 ppm F as MFP — Each subject will be randomly assigned to this treatment during one of the four periods for this crossover study.

SUMMARY:
This is a single-center, four-treatment, four-period crossover study. Over the course of the study, up to thirty qualified subjects will use four (4) study treatment products, one time each according to the randomization. Subjects will brush with 1.25g of the assigned study product at each visit. Subjects will provide saliva samples at baseline and at 2, 6, 12, and 30 minutes post-treatment. The F- concentrations in each saliva sample will be determined by ion chromatography

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent prior to study participation and be given a signed copy of the Informed Consent form;
* Be in good general health as determined by the Investigator/Designee based on a review of their medical history;
* Have at least 16 natural teeth;
* Have normal salivary flow (0.3-0.6 ml/min) or deemed acceptable by the Investigator/Designee as determined in a previous screening outside of this protocol;
* Agree not to participate in any other oral care studies for the duration of this study;
* Agree not to change their current oral care routine except 1) to refrain from using mouth rinse and 2) to agree to use study washout product as designated (current floss users are permitted to continue to floss during this study); viii. Agree to delay elective dentistry, including dental prophylaxis, until study completion, and to report any non-study dentistry received during the course of the study;
* Agree to refrain from eating, using breath mints, using medicated lozenges, chewing gum, brushing their teeth or drinking within 2 hours of the visit, other than small sips of water up to 30 minutes prior to the visit;
* Agree to refrain from drinking tea or mineral water, and/or eating sardines within the 12 hours prior to the study visit; and
* Agree to return for all scheduled visits and to follow all study procedures.

Exclusion Criteria:

* Active treatment for gingivitis, periodontitis, or caries;
* Self-reported pregnancy or nursing;
* Smoking or tobacco chewing;
* Sjögren syndrome or any other disease/condition causing severe xerostomia;
* Kidney disease or renal impairment;
* Undergoing chemotherapy or irradiation procedures;
* Fixed orthodontic appliances that may interfere with product use;
* Inability to undergo any study procedures; or
* Any condition or disease, as determined by the Investigator/Designee that could be expected to interfere with examination procedures or with the subject's safe completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
area under the curve (AUC) | 2-minutes, 6-minutes, 12-minutes, and 30-minutes
  The primary endpoint will be AUC of the fluoride levels from 2 to 30 minutes. AUC will be calculated for each subject and treatment combination by integrating a 3 parameter first order decay model curve estimate (y= theta1 * exp (-theta2.X) + theta3). For any values obtained for a timepoint that are below the detection limit, 0.5 times the detection limit will be used. The following rules will apply if a subject has missing value(s) before the AUC is calculated:
  * If 2 or more timepoints are missing within a period, then the AUC will be set to missing
  * If only 2-minute data are missing, then curve will be estimated as above
  * If 6-minute or 12-minute data are missing, a linear imputation between the adjacent timepoints will be used
  * If 30-minute data are missing, the 12-minute data will be carried forward.

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Health Science Center, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: No